CLINICAL TRIAL: NCT05890196
Title: A Pilot Study Treating Radiation Injury With Autologous Fat Transfer
Brief Title: Autologous Fat Grafting in Radiated Soft Tissue Reconstruction
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB21-1183
Record Dates: First submitted 2023-05-08; First posted 2023-06-06 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Radiation Fibrosis; Fat Grafting
MeSH Terms: conditions — Breast Neoplasms; Radiation Fibrosis Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to observe the effect of autologous fat grafting on soft tissue reconstruction of the breast following radiation treatment. Moving fat from one part of the body to another has been used for reconstruction for hundreds of years. However, it is not fully understood how well this works in reconstruction after radiation is used for cancer treatment.

DETAILED DESCRIPTION:
This is a single-arm, prospective pilot study that will objectively assess outcomes in patients electively undergoing AFT for breast or chest wall reconstruction. Patients planning to undergo autologous fat transfer for breast or chest wall reconstruction will be enrolled prospectively. As this is a pilot study, the study team plans to enroll ten (10) patients to demonstrate the feasibility of the protocol and pathway as well as establish preliminary data for extramural funding. The research will include capturing 2-dimensional (2-D) and 3-dimensional (3-D) photographs as well as ultrasound (US) soft tissue assessments to determine volume retention and changes in the reconstructed area. Participants will undergo this imaging of their breast and chest wall and complete two questionnaires to evaluate patient satisfaction, quality of life, and late effects of radiation following fat grafting over a 12-month period, all standard of care. The 3D photographs and US are routinely used in practice but will be performed for research purposes in this study.

ELIGIBILITY:
Inclusion Criteria:

* Able to give consent
* Undergoing elective autologous fat grafting
* Previously treated for breast cancer
* Previous treatment included radiation therapy to the breast/chest wall.

Exclusion Criteria:

* Unable to give consent
* No history of radiation to the breast or chest wall
* No prior treatment for breast cancer
* No indication for autologous fat grafting
* Currently pregnant or breastfeeding
* Currently consuming nicotine products (smoking, vaping, patches, gum)
* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll participants from the University of Chicago who are undergoing autologous fat grafting as part of their reconstruction for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Skin Fibrometry before and after fat transfer in reconstruction. | 12 months
  Soft tissue assessment is made using a non-invasive device SkinFibrometer (Delfin Kuopio, Finland) that measures tissue edema and skin elasticity. Measurements will be taken in all four quadrants of the affected (radiated) breast or reconstructed breast before and after the grafting procedure.

SECONDARY OUTCOMES:
Change in Radiation Injury before and after fat transfer. | 12 months
  Radiation injury assessment is made using the validated tool Late Effects Normal Tissue Task Force - Subjective Objective Management and Analytic (LENT-SOMA) score. Assessment will be made before and after the fat transfer procedure. Overall, scores are based on 12 categories, scored 0-4 with a higher score indicating more significant radiation injury.
Change in patient reported satisfaction of the breast measure before and after fat transfer. | 12 months
  The BREAST Q validated patient survey measures several realms related to breast reconstruction and allows an assessment of satisfaction and physical well-being before and after reconstruction. The survery responses are tallied and converted to a score of 100 with a higher score being more satisfied or better outcome. In addition, a change in score of 8 or more points is a clinically meaningful difference according to normative studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Summer E Hanson, Chicago, Illinois, United States

REFERENCES:
- [Background] Pattani N, Sanghera J, Langridge BJ, Frommer ML, Abu-Hanna J, Butler P. Exploring the mechanisms behind autologous lipotransfer for radiation-induced fibrosis: A systematic review. PLoS One. 2024 Jan 25;19(1):e0292013. doi: 10.1371/journal.pone.0292013. eCollection 2024. PMID 38271326
- [Background] Zheng M, Liu Z, He Y. Radiation-induced fibrosis: Mechanisms and therapeutic strategies from an immune microenvironment perspective. Immunology. 2024 Aug;172(4):533-546. doi: 10.1111/imm.13788. Epub 2024 Apr 1. PMID 38561001